CLINICAL TRIAL: NCT02407145
Title: Safety and Efficacy of Low-elasticity Polyvinylidene Fluoride (DynaMesh®-SIS Soft) Retropubic Tension Free Midurethral Sling in the Treatment of Stress Urinary Incontinence in Women
Brief Title: Safety and Efficacy of PVDF (DynaMesh®-SIS Soft) Retropubic Midurethral Slings in Stress Urinary Incontinence in Women
Status: Completed | Type: Observational
Sponsor: Julie Dawson (Other)
Collaborators: Kebomed UK (Unknown)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 2015O&G01M
Record Dates: First submitted 2015-03-24; First posted 2015-04-02 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Urinary Stress Incontinence; Urinary Incontinence,Stress
Keywords: retropubic; midurethral sling; polyvinylidene fluoride
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PVDF retropubic midurethral sling: Women with urodynamic stress urinary incontinence having a retropubic polyvinylidene fluoride midurethral sling (DynaMesh®-SIS soft).
  Interventions: Other: 24 month follow up of women with validated questionnaire

INTERVENTIONS:
Other: 24 month follow up of women with validated questionnaire — 24 month follow up (clinical and questionnaire based) of women who are already assigned to have a PVDF retropubic midurethral sling (DynaMesh®-SIS soft) as a part of their planned treatment of urodynamic stress incontinence.

SUMMARY:
This study is designed to evaluate the safety and efficacy of low elasticity polyvinylidene fluoride (DynaMesh®-SIS soft) retropubic tension-free midurethral slings in the treatment of stress urinary incontinence in women. Women who are having a retropubic PVDF midurethral sling for urodynamic stress incontinence will be followed up for 24 months to address its efficacy and rate of complications.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of low elasticity polyvinylidene fluoride (DynaMesh®-SIS soft) retropubic tension-free midurethral slings in the treatment of stress urinary incontinence (SUI) in women.

Stress urinary incontinence is a common problem, affecting large numbers of women. If conservative measures are ineffective then surgery is offered. Surgery involves a permanent mesh sling being placed, tension free beneath the midurethra. The standard retropubic tension-free vaginal tape (TVT) has been used since 1996 using a polypropylene mesh.(1) The use of permanent mesh in gynaecology has come under scrutiny due to significant complications for women.(2) This year the Medicines and Healthcare Products Regulatory Agency (MHRA), UK concluded that there is not enough evidence to withdraw mesh from clinical usage.(3)

The sling being studied is DynaMesh®SIS soft, made of polyvinylidene fluoride (PVDF) which has improved biocompatibility with tissues, meaning reduced scar formation and less mesh shrinkage.(4) Each sling is individually woven and and has low elasticity meaning dimensions are maintained under tension, such as with coughing or straining. The technique of retropubic placement of the DynaMesh®SIS soft does not differ from current retropubic TVT placement.

The hypothesis is that the low elasticity polyvinylidene fluoride midurethral sling is non-inferior in both safety and efficacy compared with the safety and efficacy of traditional polypropylene slings, as reported in current literature.

There are eleven research centres in two countries, The United Kingdom and Ireland. The DynaMesh®SIS soft sling is currently in use in four of eleven of the research hospitals, Norwich (main research centre), Antrim and Belfast in the UK and in Munich in Germany. It will be introduced in London, Cambridge, Wirral, Solihull, Huntingdon and Kilmarnock in the UK and Wurzbug in Germany.

Women with urodynamic stress incontinence who are already assigned to have this retropubic midurethral tape placed for treatment will be recruited prior to their procedure for ongoing follow up. Participants will complete standardised urinary incontinence and quality of life questionnaires prior to their procedure and at 3,6,12, 18 and 24 months by post. Clinical follow up will occur at 3 and 12 months post operatively and as required if any concerns.

ELIGIBILITY:
Inclusion Criteria:

* women with proven urodynamic stress incontinence in whom a retropubic midurethral sling is appropriate treatment as per the treating urogynaecologist, gynaecologist or urologist
* women who have not had a previous incontinence procedure
* no concomitant prolapse procedure at the time of sling placement

Exclusion Criteria:

* urodynamic studies negative for stress urinary incontinence
* previous incontinence procedures
* non English/non German speaker depending on study centre
* lack capacity to consent

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women presenting with urinary incontinence, presenting to the research centres through normal referral pathways
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The subjective cure rate of retropubic midurethral PVDF slings in treating stress urinary incontinence. | 3 to 24 months
The rate of complications of retropubic midurethral PVDF slings, in particular mesh erosions. | 3 to 24 months

SECONDARY OUTCOMES:
Changes in quality of life, with regards to urinary symptoms, following placement of a retropubic midurethral PVDF sling. | 3 to 24 months
The subjective cure rate of retropubic midurethral PVDF slings in treating stress urinary incontinence compared to the reported cure rate for traditional polypropylene retropubic slings. | 3 to 24 months
The rate of complications of retropubic midurethral PVDF slings, in particular vaginal erosions and how the rates of complications compare to those reported in the literature for traditional polypropylene retropubic slings. | 3-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sambit Mukhopadhyay, Principal Investigator — Norfolk and Norwich University Hospital Trust; Edward P Morris, Study Chair — Norfolk and Norwich University Hospital Trust
Locations (10):
- Germany (2):
  - Chirurgische Klinik, Munich
  - Universitätsklinikum Würzburg, Würzburg
- United Kingdom (8):
  - Hichingbooke Hospital, Huntingdon, Cambridgeshire
  - Addenbrooke's Hospital, Cambridge, Cambrigeshire
  - South Eastern Health and Social Care Trust, Belfast
  - NHS Ayrshire & Arran, Kilmarnock
  - University College Hospital, London
  - Wirral University Teaching Hospital NHS Foundation, Metropolitan Borough of Wirral
  - Norfolk and Norwich University Hospitals Trust, Norwich
  - Heart of England NHS Foundation Trust, Solihull

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ulmsten U, Henriksson L, Johnson P, Varhos G. An ambulatory surgical procedure under local anesthesia for treatment of female urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):81-5; discussion 85-6. doi: 10.1007/BF01902378. PMID 8798092
- [Background] U.S. FDA Safety Communication: urogynecologic surgical mesh: update on the safety and effectiveness of transvaginal placement for pelvic organ prolapse. July 2011
- [Background] A summary of the evidence on the benefits and risks of vaginal mesh implants. October 2014. Medicines and Healthcare Products Regulatory Agency, United Kingdom.
- [Background] Klinge U, Binneboesel M, Kuschel S, Schuessler B. Demands and properties of alloplastic implants for the treatment of stress urinary incontinence. Expert Rev Med Devices. 2007 May;4(3):349-59. doi: 10.1586/17434440.4.3.349. PMID 17488229

DOCUMENTS (2):
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT02407145/Prot_000.pdf
  • Informed Consent Form (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT02407145/ICF_001.pdf